CLINICAL TRIAL: NCT01863836
Title: Randomized Trial of Fluoroscopy Use for Radial Endobronchial Ultrasound-guided Biopsy of Peripheral Lung Lesions
Brief Title: Study on the Influence of Fluoroscopy in the Diagnosis of Peripheral Lung Lesions With Endobronchial Ultrasound Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Responsible Party: Principal Investigator, Antoine Delage, MD, Laval University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IUCPQ-20913
Record Dates: First submitted 2013-04-19; First posted 2013-05-29 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-09

CONDITIONS: Peripheral Pulmonary Lesions
Keywords: Radial endobronchial ultrasound; Peripheral lung lesion; Fluoroscopy; Lung cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fluoroscopy (Experimental): Patients will undergo bronchoscopy and radial endobronchial ultrasound-guided biopsy of a peripheral lung lesion like patients in the other group. However, single-plane fluoroscopy will be used to help locate the lesion (with the help of a steerable curette) in case of failure to locate the lesion, and it will also be used to guide tissue sampling and ensure appropriate sampling tool function. Transbronchial biopsies, transbronchial needle aspiration, brushings, and bronchoalveolar lavage will be performed for each lesion.
  Interventions: Procedure: Fluoroscopy; Procedure: Radial EBUS-guided biopsy
- No fluoroscopy (Active Comparator): Patients will undergo biopsy of peripheral lung lesions using radial endobronchial ultrasound guidance only, without the use of fluoroscopy. Transbronchial biopsies, transbronchial needle aspiration, brushings, and bronchoalveolar lavage will be performed for each lesion.
  Interventions: Procedure: Radial EBUS-guided biopsy

INTERVENTIONS:
Procedure: Fluoroscopy
  Arms: Fluoroscopy
Procedure: Radial EBUS-guided biopsy

SUMMARY:
The purpose of this study is to determine whether the use of fluoroscopy improves the diagnostic yield of peripheral pulmonary lesions' biopsy guided by radial endobronchial ultrasound (with the use of a guide sheath).

DETAILED DESCRIPTION:
See above

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients referred for the bronchoscopic diagnosis of peripheral pulmonary lesions at the Institut Universitaire de Cardiologie et de Pneumologie de Québec(not visible endobronchially)
* Adults over the age of 18

Exclusion Criteria:

* Therapeutic anticoagulation
* Antiplatelet therapy other than aspirin
* Known hemorrhagic diathesis
* Acute respiratory failure
* Pregnancy
* Inability to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2013-04; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Diagnostic yield | Upon production of pathology results, usually within 2 weeks after the test
  Diagnostic yield of radial endobronchial ultrasound-guided biopsy for peripheral lung lesions defined as the proportion of patients in whom a specific diagnosis is established by radial endobronchial ultrasound-guided biopsy. The analysis will be stratified by lesion size, location, the presence of the bronchus sign, type of echographic image obtained (central/peripheral), physician involved, resident involvement.
Sensitivity and specificity | Upon completion of ancillary or confirmatory tests, usually within 2 months after the test
  Sensitivity and specificity are determined separately for malignancy and benign etiologies. Case records will be reviewed for patients with non-diagnostic specimen and results from other diagnostic procedures (TTNA, surgical biopsy) will be reviewed. For patients without further diagnostic tests, stability or progression of the lesion over time will be used for etiology attribution.

SECONDARY OUTCOMES:
Lesion localization | Immediate (during the test)
  Proportion of patients in whom the peripheral pulmonary lesion was localized using the radial endobronchial ultrasound.
Procedure duration | During the test
  Total duration of the bronchoscopic test.
Complications | Immediately during the test and up to 4 hours after the test
  occurrence of pneumothorax (and its management), bleeding more than 50ml, sustained desaturation below 90%, cardiac dysrhythmias, or any other adverse events occuring during or after the procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Antoine Delage, MD, Principal Investigator — Institut universitaire de cardiologie et de pneumologie de Québec, University Laval
Locations (1):
- Institut Universitaire de Cardiologie et de Pneumologie de Québec, Université Laval, Québec, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No